CLINICAL TRIAL: NCT01791738
Title: Comparison of Acetabular Shell Position Using Patient Specific Instruments vs. Standard Surgical Instruments: A Randomized Clinical Trial
Brief Title: Acetabular Shell Positioning Using Patient Specific Instruments
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Wael Barsoum, Vice Chairman , Orthpaedic Surgery, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCF 10-1138
Record Dates: First submitted 2013-02-07; First posted 2013-02-15 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Osteoarthritis, Hip; Rheumatoid Arthritis; Avascular Necrosis
Keywords: Total Hip Arthroplasty (THA); Patient-Specific Instruments; Acetabular Cup Placement; Accuracy
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis, Rheumatoid; Osteonecrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetabular positioning system (Experimental): Pre-operative planning through 3D software with design and fabrication of patient specific instruments for placement of a guide pin to be used to aid in bone preparation for insertion of an acetabular cup in total hip arthroplasty
  Interventions: Procedure: Acetabular positioning system
- Standard total hip arthroplasty (No Intervention): Each surgeon will use their standard methods of pre-operative planning using pre-operative x-rays, and complete the procedure using standard surgical instruments for total hip arthroplasty.

INTERVENTIONS:
Procedure: Acetabular positioning system — Pre-operative planning through 3D software with design and fabrication of patient specific instruments for placement of a guide pin to be used to aid in bone preparation for insertion of an acetabular cup in total hip arthroplasty
  Arms: Acetabular positioning system

SUMMARY:
The proposed study is a double-blinded randomized controlled trial comparing patient specific instruments with solely standardized instruments and pre-operative planning used for the placement of the acetabular cup prosthesis used in total hip arthroplasty.

The investigators will enroll 36 patients who have consented to total hip arthroplasty for treatment of hip pathology. This treatment is a standard of care. Patients will receive standard of care pre- and post-operative care and placement of standard of care implants all of which are commercially available and FDA approved for general use for the clinical indications used in these patients. All patients will receive a pre-operative CT scan for surgical planning and comparison with post-operative CT scan. The difference in intervention between the groups will be the creation and use of patient specific instruments from the pre-operative planning session. These instruments will be used for placement of an indexing peripheral guide wire to direct acetabular preparation and placement of the shell assisting standard surgical instruments. Print-offs from the pre-operative plan will also be used in the treatment group.

The post-operative scan will be performed within two weeks of the surgery for both the treatment and control groups. The investigators will analyze the difference in acetabular shell placement (acetabular version and abduction angle) from the pre-operatively planned CT scan. These differences will be compared between the control and experimental groups.

DETAILED DESCRIPTION:
No further details to report.

ELIGIBILITY:
Inclusion Criteria:

Subjects to be included in this protocol will be adult males and females of all races and socioeconomic status meeting the following criteria:

* Primary, unilateral direct lateral or posterior THA
* 18 to 85 years old at time of surgery
* Able to get a pre- and post-operative CT scan at the Cleveland Clinic

Exclusion Criteria:

* The following criteria will exclude subjects from this protocol:
* Significant metal in the joint that results in metal artifact on the pre--operative CT scan, thereby compromising the ability to visualize the acetabulum on the pre-operative simulator.
* Pregnancy
* Incarceration
* Condition deemed by physician or medical staff to be non-conducive to patient's ability to complete the study, or a potential risk to the patient's health and well-being.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Difference between planned and actual values of Abduction and Version. | Through 2 weeks after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Wael K Barsoum, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States